CLINICAL TRIAL: NCT04598932
Title: Corneal Biomechanical Analysis Using Brillouin Microscopy
Status: Enrolling by invitation | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: University of Maryland (Other)
Responsible Party: Principal Investigator, James Bradley Randleman, Staff Physician, The Cleveland Clinic
Other Study IDs: 20-355
Record Dates: First submitted 2020-05-19; First posted 2020-10-22 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-09

CONDITIONS: Keratoconus; Keratoconus, Unstable; Keratoconus, Stable
Keywords: Brillouin; Keratoconus; Keratoconus, Unstable; Corneal Cross Linking; CXL; LASIK; PRK; SMILE
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (6):
- 1: Normal Controls: Patients with normal corneas without any prior surgery to serve as the control group
  Interventions: Device: Brillouin microscopy
- 2 Keratoconus: Patients with various stages of keratoconus
  Interventions: Device: Brillouin microscopy
- 3: LASIK: Patients with normal corneas who are undergoing laser in situ keratomileusis (LASIK)
  Interventions: Device: Brillouin microscopy
- Group 4: PRK: Patients with normal corneas who are undergoing photorefractive keratectomy (PRK)
  Interventions: Device: Brillouin microscopy
- 5: SMILE: Patients with normal corneas who are undergoing small incision lenticular extraction (SMILE)
  Interventions: Device: Brillouin microscopy
- 6: CXL: Patients with keratoconus who are undergoing corneal cross-linking (CXL)
  Interventions: Device: Brillouin microscopy

INTERVENTIONS:
Device: Brillouin microscopy — The Brillouin clinical instrument is comprised of three parts: a human interface, a laser-scanning confocal microscope, and an etalon-based spectrometer. The human interface is a modified ophthalmic slit-lamp instrument with chin support and headrest. The light source is a single longitudinal mode CW laser at 780 nm. A polarizing beam splitter and quarter-wave plate assembly sends the laser beam to the human interface. To focus light into the eye, a long-working distance microscope objective is used. Brillouin scattered light from the eye is collected with a single-mode optical fiber. For spectral analysis, a two-stage VIPA-etalon spectrometer configured with the cross-axis cascade principle and the spectrum is measured on a EM-CCD camera.

SUMMARY:
The objective of this study is to measure the Brillouin biomechanical properties in keratoconic corneas and characterize biomechanical alterations that occur after corneal procedures that inherently strengthen or weaken the cornea by evaluating the change in Brillouin metrics before and after treatments.

DETAILED DESCRIPTION:
Surgical correction of myopia and keratoconus identification/management are separate but tightly intertwined issues of major significance. For both, there is an unmet need for direct measurements to evaluate corneal stiffness (i.e. its resistance to deformation). The prevalence of myopia is expected to double, affecting more than 50% of the US population, by 2050. Laser in situ keratomileusis (LASIK) is one of the most popular and successful surgeries in the world and compares favorably to long-term contact lens wear use for myopia correction. However, only ~10% of eligible patients undergo LASIK currently; the others cite safety concerns as a major factor in their decision. The primary risk for poor refractive surgery outcomes is biomechanical failure due to unidentified (subclinical) ectasia (i.e. keratoconus). Patients presenting for LASIK evaluation with atypical, suspicious corneal curvature but with undetermined true risk represent the leading reason for surgery screening failures. This results in good candidates being denied surgery, while up to 10% of truly poor candidates are still missed using current screening algorithms.

Keratoconus is up to 10 times more prevalent than the previously reported 1/2000 figure. Corneal cross-linking (CXL) is now FDA approved in the US for keratoconus treatment and is effective at stiffening the cornea and halting ectasia progression. Early identification of keratoconus is critical, but current tests in the clinic are morphological, not biomechanical, and therefore do not allow a definitive diagnosis at the earliest stages resulting in vision loss before CXL treatment is initiated. Thus, the need for accurate identification of subclinical ectasia has never been greater.

In the past years, newly developed technology, Brillouin microscopy, has emerged as the most promising tool to address this clinical need. This study will systemically address the critical gap in current knowledge by linking Brillouin mapping of corneal biomechanical alterations to abnormal morphological behavior and testing the findings in conditions where corneal biomechanics are abruptly altered, by: 1) weakening with refractive surgery procedures, and 2) strengthening through corneal cross-linking.

It is anticipated that a clinical tool assessing the mechanical state of the cornea will improve early diagnosis and management of keratoconus as well as refractive surgery planning. Ultimately, this will lead to predictive models where Brillouin measurements could be an accurate predictor of postoperative outcomes and thus aid in developing individualized surgical parameters.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-60 with keratoconus
* patients aged 18-60 with normal corneas,
* patients aged 18-60 undergoing refractive surgery (LASIK, PRK, SMILE)
* patients aged 18-60 with keratoconus undergoing CXL

Exclusion Criteria:

* outside age range
* history of previous ocular surgeries
* unable to cooperate for the Brillouin microscopic examination
* unable to provide informed consent

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Group 1: Patients with normal corneas Group 2: Patients with keratoconus Group 3: Patients with normal corneas undergoing LASIK Group 4: Patients with normal corneas undergoing PRK Group 5: Patients with normal corneas undergoing SMILE Group 6: Patients with keratoconus undergoing CXL
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Brillouin Metrics | Difference between baseline and 3 months after intervention
  Brillouin metrics to be evaluated include localized Mean Brillouin modulus measure across the cornea and at each depth of the corneal stroma

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Cole Eye Institute, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
there is no plan to share data

REFERENCES:
- [Background] Zhang H, Roozbahani M, Piccinini AL, Golan O, Hafezi F, Scarcelli G, Randleman JB. Depth-Dependent Reduction of Biomechanical Efficacy of Contact Lens-Assisted Corneal Cross-linking Analyzed by Brillouin Microscopy. J Refract Surg. 2019 Nov 1;35(11):721-728. doi: 10.3928/1081597X-20191004-01. PMID 31710374
- [Background] Webb JN, Langille E, Hafezi F, Randleman JB, Scarcelli G. Biomechanical Impact of Localized Corneal Cross-linking Beyond the Irradiated Treatment Area. J Refract Surg. 2019 Apr 1;35(4):253-260. doi: 10.3928/1081597X-20190304-01. PMID 30984983
- [Background] Randleman JB, Su JP, Scarcelli G. Biomechanical Changes After LASIK Flap Creation Combined With Rapid Cross-Linking Measured With Brillouin Microscopy. J Refract Surg. 2017 Jun 1;33(6):408-414. doi: 10.3928/1081597X-20170421-01. PMID 28586502
- [Result] Scarcelli G, Pineda R, Yun SH. Brillouin optical microscopy for corneal biomechanics. Invest Ophthalmol Vis Sci. 2012 Jan 20;53(1):185-90. doi: 10.1167/iovs.11-8281. PMID 22159012
- [Result] Scarcelli G, Kling S, Quijano E, Pineda R, Marcos S, Yun SH. Brillouin microscopy of collagen crosslinking: noncontact depth-dependent analysis of corneal elastic modulus. Invest Ophthalmol Vis Sci. 2013 Feb 19;54(2):1418-25. doi: 10.1167/iovs.12-11387. PMID 23361513
- [Result] Scarcelli G, Besner S, Pineda R, Yun SH. Biomechanical characterization of keratoconus corneas ex vivo with Brillouin microscopy. Invest Ophthalmol Vis Sci. 2014 Jun 17;55(7):4490-5. doi: 10.1167/iovs.14-14450. PMID 24938517
- [Result] Scarcelli G, Besner S, Pineda R, Kalout P, Yun SH. In vivo biomechanical mapping of normal and keratoconus corneas. JAMA Ophthalmol. 2015 Apr;133(4):480-2. doi: 10.1001/jamaophthalmol.2014.5641. No abstract available. PMID 25611213